CLINICAL TRIAL: NCT03868904
Title: OCS Lung INSPIRE Long-Term Continuation Post-Approval Study - INSPIRE Continuation PAS
Brief Title: INSPIRE Continuation Post-Approval Study
Status: Completed | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LUN-03-PAS
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-11

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- OCS Lung INSPIRE Trial
  Interventions: Device: OCS Lung System

INTERVENTIONS:
Device: OCS Lung System — No active interventions are part of this study. This study will collect long-term survival and BOS data in subjects who were part of the INSPIRE trial.

SUMMARY:
To evaluate long-term BOS-free survival outcomes of the OCS™ Lung INSPIRE Trial patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant in TransMedics OCS Lung System INSPIRE trial

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who participated in TransMedics OCS Lung System INSPIRE Trial
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Brochiolitis Obliterans Syndrome (BOS) -free survival | 5 years post transplant
  BOS-free survival

SECONDARY OUTCOMES:
Survival | 5 years
  Survival post transplant
Freedom from Bronchiolitis Obliterans Syndrome (BOS) as determined from pulmonary function tests (PFT's) | 5 years
  Freedom from BOS

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- St. Vincent's Hospital, Darlinghurst, New South Wales, Australia
- University of Leuven Hospital, Leuven, Belgium
- University of Alberta, Edmonton, Alberta, Canada
- N.H.C Hospital Civil, Strasbourg, France
- Germany (2):
  - German Heart Institute Berlin, Berlin
  - Hannover Medical School, Hanover
- University of Padua, Padua, Italy
- Hospital Universitario Puerta De Hierro, Madrid, Spain
- United Kingdom (2):
  - Papworth Hospital, Cambridge
  - Harefield Hospital, Middlesex

IPD SHARING:
Plan to Share IPD: No